CLINICAL TRIAL: NCT02437526
Title: Analytic Treatment Interruption of Antiretroviral Therapy to Assess for HIV Cure
Brief Title: Analytic Treatment Interruption (ATI) to Assess HIV Cure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andrew D. Badley, M.D., Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-001678
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: HIV
Keywords: Cure; Analytic treatment interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment interruption (Experimental): Antiretroviral therapy will be discontinued under close laboratory monitoring and clinical supervision.
  Interventions: Other: Analytic treatment interruption

INTERVENTIONS:
Other: Analytic treatment interruption

SUMMARY:
This study is designed to determine if individual patients with HIV infection have been cured of the infection. To do this, antiretroviral therapy is discontinued under close medical supervision and the patient monitored over time for reactivation of infection.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* HIV-1 infected with the potential to have been cured of infection in the course of routine clinical care in the opinion of the treating physician and study team
* Have an undetectable plasma HIV-1 RNA and undetectable proviral DNA on suppressive antiretroviral therapy on at least two consecutive measures for at least 6 months
* Able and willing to either abstain from sexual activity or use barrier contraceptives during the ATI
* Negative serum β-HCG pregnancy test in women with childbearing potential
* Have the ability to give appropriate informed consent.

Exclusion Criteria

* Women who are pregnant or nursing
* Women who can become pregnant who are unable or unwilling to use both barrier and pharmacologic contraceptives during the ATI
* Previous or current infections that are at high risk of reactivating with immune suppression, in whom there are no effective antimicrobial prophylaxis options
* Advanced cardiopulmonary or liver disease
* History of untreated solid or hematologic malignancies
* Evidence of active viral replication in patients co-infected with Hepatitis B virus (HBV). Treatment should be provided to suppress HBV replication with agents that do not have activity against HIV (ie entecavir) prior to consideration for ATI.
* Evidence of viral replication with Hepatitis C virus (HCV), together with evidence of any hepatic fibrosis or inflammation. Such patients should be offered HCV treatment first.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-05; Primary Completion 2035-05 (Estimated); Study Completion 2035-05 (Estimated)

PRIMARY OUTCOMES:
Time to virologic rebound | 38 weeks

SECONDARY OUTCOMES:
Time to HIV-1 RNA ≥ 20 copies/ml | 38 weeks
Time to HIV-1 RNA ≥ 100 copies/ml | 38 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Badley, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials